CLINICAL TRIAL: NCT05659745
Title: Randomized, Double-blind, Placebo-controlled Trial Investigating the Role of a Personal Care Product on Vaginal Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seed Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 20259
Record Dates: First submitted 2022-12-01; First posted 2022-12-21 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-01

CONDITIONS: Vaginal Personal Care
Keywords: Lactobacillus crispatus; vaginal odor; vaginal health

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Due to this study being double-blind, participants will not know if they are in the condition with the test product or the placebo. Neither the test products nor the placebo used during the study will be labeled in any way that will indicate whether participants are taking the placebo or the test product. Participants will just know there is a chance they were randomized into a placebo or test product arm of the study. As mentioned above, only the Research Coordinator will know which group the participant is randomized into. The PI will remain blinded throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Vaginal Suppository Capsule (Placebo Comparator): In the VM-02 Vaginal Suppository Capsule Placebo Arm, participants will take the test vaginal suppository capsule placebo as directed.
  Interventions: Other: VM-02 Placebo
- Vaginal Suppository Capsule Active (Experimental): In the VM-02 Vaginal Suppository Capsule Active Arm, participants will take a test vaginal suppository capsule as directed.
  Interventions: Other: VM-02
- Vaginal Suppository Tablet Active (Experimental): In the VM-02 Vaginal Suppository Tablet Active Arm, participants will take a test vaginal suppository tablet as directed.
  Interventions: Other: VM-02
- Oral Capsule Active (Experimental): In the VM-02 Oral Capsule Active Arm, participants will take a test oral capsule as directed.
  Interventions: Other: VM-02
- Commercial Oral Vaginal Probiotic Competitor (Other): In the Commercial Over-The-Counter (OTC) Oral Probiotic Competitor Arm, participants will take an over-the-counter competitor product as directed.
  Interventions: Dietary Supplement: Commercial Oral Probiotic Competitor

INTERVENTIONS:
Other: VM-02 — VM-02 is a personal care product for vaginal health.
  Arms: Oral Capsule Active; Vaginal Suppository Capsule Active; Vaginal Suppository Tablet Active
Dietary Supplement: Commercial Oral Probiotic Competitor — Commercial Oral Vaginal Probiotic Competitor is a personal care product for vaginal health.
  Arms: Commercial Oral Vaginal Probiotic Competitor
Other: VM-02 Placebo — VM-02 Placebo is a personal care product placebo for vaginal health.
  Arms: Vaginal Suppository Capsule

SUMMARY:
The goal of this clinical trial is to assess the impact of a personal care product on vaginal health in a healthy participant population. The personal care product, VM-02, contains a prebiotic, postbiotic, and three distinct strains of Lactobacillus crispatus, a microbe commonly found in healthy females, together accounting for greater than 85% of known genes in this species. The intervention will be compared to a placebo intervention and will aim to assess the following in a healthy female population:

Measure changes in the relative and absolute abundance of a bacterial species, Lactobacillus crispatus, in the vagina, compared the baseline (prior to use of the personal care product) to two time points after use.

Observe changes in vaginal pH and self-reported discomfort from vaginal odor, compared the baseline to two time points after use.

Determine the user experience of three variations of a personal care product administered in different formats to improve vaginal health and establish tolerability and user acceptability.

Participants will use the personal care product according to a specific program as directed, conduct vaginal swab sampling, and answer questionnaires, each at eight time points.

DETAILED DESCRIPTION:
The vaginal microbiome is a dynamic microecosystem that undergoes fluctuations during the female menstrual cycle and at various life stages from puberty to menopause. A healthy vaginal microbiome is dominated by Lactobacillus which regulates vaginal pH, produces antimicrobial compounds, and significantly influences host immune response. The purpose of this study is to determine whether vaginal health can be influenced by a novel personal care product comprised of a Lactobacillus postbiotic, prebiotic, and multiple strains of Lactobacillus crispatus predictive of a stable vaginal microbiome.

This study will be a randomized double-blind, placebo-controlled intervention that will examine the safety and tolerability of a personal care product for vaginal health, VM-02. This pilot study will last for the duration of two complete menstrual cycles. Data will be collected via participant virtual questionnaires and vaginal swabs.

Participants are randomized as follows:

A two-arm randomized, double-blind, placebo-controlled study to evaluate VM-02 as a vaginal suppository capsule.

Arm #1: Vaginal application of single-use applicators filled with a vaginal suppository capsule at 5 x 10^8 CFU/dose. The study product will be administered once daily for 7 consecutive days, followed by once weekly application over 2 consecutive additional weeks.

Arm #2: Vaginal application of single-use applicators filled with a vaginal suppository placebo capsule. The study product will be administered once daily for 7 consecutive days, followed by once weekly application over 2 consecutive additional weeks.

Three additional arms are included to quantify the impact of an alternative formulation and user experience.

Arm #3: Vaginal application of single-use applicators filled with vaginal suppository tablet at 5 x 10^8 CFU/dose. The study product will be administered on Days 1,4,7,14,21.

Arm #4: Oral administration of capsule at 5 x 10^8 cfu/dose. The study product will be administered daily for 30 consecutive days.

Arm #5: Oral administration of commercially available over-the-counter oral capsule at 5 x 10^8 CFU/dose. The study product will be administered daily for 30 consecutive days.

Colonization rate of 3 distinct Lactobacillus crispatus after administration of VM-02 will be assessed with PCR and DNA sequence analysis.

Researchers will compare groups who received active product with those who received a placebo (a look-alike substance that contains no active drug) to determine product safety and any possible side effects, see if the amount of the bacterial species, Lactobacillus crispatus, changes (either increases or decreases) in response to the treatment, and to determine any impacts on self-reported odor and vaginal health.

A total of 80 participants will be recruited for this study. All participants will be supported and tracked through the various stages of the study virtually. All biomarker swabs that are taken by participants will be returned via pre-paid envelopes provided by the research team and all survey information will be collected online. No in-person visits will be required. Participants who are unwilling to follow the study protocol will be removed from the study.

ELIGIBILITY:
Inclusion Criteria:

* Reproductive age women aged ≥ 18.
* History of regular menses every 21-35 days for six months prior to the study.
* Agreement not to use specified intra-vaginal products during the study product use.
* Willing to use an intra-vaginal suppository or dietary supplement during the study period.
* Willing to complete vaginal swabs on themselves as directed in the study.
* Ability to understand and read English and provide written consent.

Exclusion Criteria:

* Pregnancy or planned pregnancy in the next 6 months.
* Two or more amenorrheic months in the past 6 months.
* Lives in the state of New York.
* Allergy to any components of the supporting or excipient ingredients in test formulation capsules, tablets, placebos or over-the-counter competitor product.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of VM-02 at 5 x 10^8 CFU/dose based on frequency and absolute number of patient reported adverse events | Throughout intervention and subsequent 4 week period following last dose

SECONDARY OUTCOMES:
Vaginal colonization calculated by detection of each of 3 distinct Lactobacillus crispatus strains after administration of VM-02 at 5 x 10^8 CFU/dose using metagenomic sequencing and/or strain-specific PCR-based assays | 2 and 4 weeks after intervention

OTHER OUTCOMES:
Self-reported pH values after administration of VM-02 at 5 x 10^8 CFU/dose | 2 and 4 weeks after intervention
Cytokine panel assays after administration of VM-02 at 5 x 10^8 CFU/dose | 2 and 4 weeks after intervention
Participant self-reported questionnaire outcomes after administration of VM-02 at 5 x 10^8 CFU/dose | 2 and 4 weeks after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Seed Health, Venice, California, United States

REFERENCES:
- [Derived] Ravel J, Simmons S, Jaswa EG, Gottfried S, Greene M, Kellogg-Spadt S, Gevers D, Harper DM. Impact of a multi-strain L. crispatus-based vaginal synbiotic on the vaginal microbiome: a randomized placebo-controlled trial. NPJ Biofilms Microbiomes. 2025 Aug 9;11(1):158. doi: 10.1038/s41522-025-00788-6. PMID 40783570
- See also: Related Info — http://www.seedhealth.com